CLINICAL TRIAL: NCT01762241
Title: Xbox Kinect Training in Men With Metastatic Prostate Cancer Receiving Androgen Deprivation Therapy
Brief Title: Xbox Kinect Training in Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitalsenheden Vest (Other)
Responsible Party: Principal Investigator, Brigitta R. Villumsen, PhD stud., Study Nurse, Master of Science in Nursing, Hospitalsenheden Vest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wii-1-10-72-593-12; 1-10-72-593-12 (Other: Hospitalsenheden Vest)
Record Dates: First submitted 2012-12-20; First posted 2013-01-07 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Androgen deprivation therapy; Exercise; Xbox
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): 12 weeks systematically home based training 3 times per week one hour at the time using the Xbox Kinect system.
  Interventions: Behavioral: Home based training using the Xbox Kinect system
- Control group (No Intervention): No systematically training/standard of care

INTERVENTIONS:
Behavioral: Home based training using the Xbox Kinect system — Home based training 3 times a week for 12 weeks using the Xbox Kinect system
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the effect of 12 weeks systematically training using the Xbox Kinect system.

Outcome measures are made on physical function, quality of life, fatigue and metabolic parameters.

DETAILED DESCRIPTION:
Patients will be recruited from the outpatient clinic at the urological department, Regionshospitalet Holstebro.

Patients who have been discharged from the outpatient clinic due to biochemical stabile cancer prostate disease will receive a letter with information about the study.

A research assistant will be responsible for randomization and test procedures. A physiotherapist will be responsible for instruction of the participants to the training and the Xbox system.

A student will be responsible for installation and collection of the Xbox system in the participants home.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer requiring androgen deprivation therapy
* Androgen deprivation therapy for at least 3 month prior to inclusion
* Cognitive well-functioning in order to be able to answer questionnaires and train according to instructions
* Signed informed consent

Exclusion Criteria:

* Prostate cancer with metastasis to other regions than bones
* Strength- or cardiovascular training 2 times or more per week prior to inclusion
* Haemoglobin percentage less than 6,1 mmol/l
* Any mental or physical condition that makes the patient unfit for participation
* Men in risk of getting an osteoporotic fracture due to long-term treatment with steroids or earlier fractures due to minimal trauma
* Participation in other studies

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The effect of 12 weeks systematically training with the Xbox Kinect system on physical function | Change from baseline to week 12
  6 min walk test

SECONDARY OUTCOMES:
The effect of 12 weeks systematically training with the Xbox Kinect on body composition | Change from baseline to week 12
  Method: BIoelectrical impedance analysis Bioelectrical impedance
The effect of 12 weeks systematically training with the Xbox Kinect system on physical function | Change from baseline to week 12
  Leg extensor power
The effect of 12 weeks systematically training with the Xbox Kinect system on fatigue | Change from baseline to week 12
  Fatigue measured using the Functional Assessment of Canter Therapy-Fatigue questionnaire
The effect of 12 weeks systematically training with the Xbox Kinect system on quality of life | Change from baseline to week 12
  Quality of life measured using the Functional Assessment of Canter Therapy-Prostate questionnaire
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12
  Waist circumference (cm)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12
  Blood pressure (mmHg)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12
  Body weight (kg)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Blood glucose (mmol/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Plasma triglyceride (mmol/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Plasma cholesterol (mmol/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Plasma High-density lipoprotein (HDL-cholesterol) (mmol/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Plasma Low-density lipoprotein (LDL-cholesterol) (mmol/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Leptin (µg/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Adiponectin (mg/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on metabolic parameters | Change from baseline to week 12 and week 24
  Leptin:Adiponectin ratio
The effect of 12 weeks systematically training with the Xbox Kinect system on the prevalence of the metabolic syndrome | Change from baseline to week 12
  The five components of the metabolic syndrome: blood glucose, triglyceride, HDL-cholesterol, waist circumference, blood pressure
The effect of 12 weeks systematically training with the Xbox Kinect system on insulin | Change from baseline to week 12 and week 24
  Insulin (pmol/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on insulin resistance | Change from baseline to week 12 and week 24
  Homeostasis model assessment for insulin resistance (HOMA-IR)
The effect of 12 weeks systematically training with the Xbox Kinect system on Insulin Growth Factor-I (IGF-I), bioactive IGF, and IGF-II | Change from baseline to week 12 and week 24
  IGF-I, bioactive IGF and IGF-II (µg/L)
The effect of 12 weeks systematically training with the Xbox Kinect system on Insulin Growth Factor Binding Protein 1-3 (IGFBP 1-3) | Change from baseline to week 12 and week 24
  IGFBP 1-3 (µg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta R Villumsen, M.S.N., Principal Investigator — Hospitalsenheden Vest
Locations (3):
- Denmark (3):
  - Urinvejskirurgisk afdeling, Aarhus Universitetshospital, Skejby, Aarhus
  - Regionshospitalet Holstebro, Urinvejskirurgisk afdeling, Holstebro
  - Urologisk afdeling, Regionshospitalet Viborg, Viborg